CLINICAL TRIAL: NCT01129791
Title: Comparison of Raw Milk Consumption vs. Other Milk Sources on Lactose Digestion in Healthy Individuals With Self-reported Lactose Intolerance
Brief Title: Effects of Raw Versus Other Milk Sources on Lactose Digestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Christopher Gardner, Professor of Medicine (Research), Stanford University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SU-05062010-5882
Record Dates: First submitted 2010-05-21; First posted 2010-05-25 (Estimated); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Lactose Intolerance
Keywords: Lactose intolerance; Dairy products; Raw milk; Adults
MeSH Terms: conditions — Lactose Intolerance | interventions — Milk

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Raw Milk first (Experimental): Organic raw cow's milk
  Interventions: Behavioral: Raw Milk
- Pasteurized milk first (Placebo Comparator): Organic pasteurized cow's milk
  Interventions: Behavioral: Pasteurized Milk
- Non-Dairy Milk first (Placebo Comparator): Unflavored soy milk
  Interventions: Behavioral: Non-dairy milk

INTERVENTIONS:
Behavioral: Raw Milk — Organic whole raw cow's milk, consumed daily in one sitting, at incremental doses from 4 to 24 oz. for 8 days. After a 1-week wash-out period, pasteurized cow's milk or non-dairy milk were consumed in the same fashion for another 8 days each.
  Arms: Raw Milk first
Behavioral: Pasteurized Milk — Organic whole pasteurized cow's milk, consumed daily in one sitting, at incremental doses from 4 to 24 oz. After a 1-week wash-out period, raw cow's milk or non-dairy milk were consumed in the same fashion for another 8 days each.
  Arms: Pasteurized milk first
Behavioral: Non-dairy milk — Unflavored soy milk, consumed daily in one sitting, at incremental doses from 4 to 24 oz. After a 1-week wash-out period, raw cow's milk or pasteurized cow's milk were consumed in the same fashion for another 8 days each.
  Arms: Non-Dairy Milk first

SUMMARY:
The purpose of this small, short pilot study is to determine the feasibility (e.g., recruitment, dose acceptance, retention) of a future longer trial comparing the effects of different types of milk (raw milk, cow's milk, nondairy-milk) on lactose maldigestion.

DETAILED DESCRIPTION:
The goal is to determine if raw milk consumption intake will benefit humans with lactose maldigestion, a common human response to the intake of dairy products during adult years. An increasing number of people are consuming raw unpasteurized milk. Enhanced nutritional qualities, taste, and health benefits have all been advocated as reasons for increased interest in raw milk consumption.

However, science-based data to substantiate these claims are limited or anecdotal.

Raw milk may differ in its ability to improve lactose maldigestion related symptoms from other milk types. Adult lactose maldigestion affects the majority of the world adult population. It appears that consumption of lactose containing foods by those who cannot digest lactose is a relatively common cause of irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Both women and men
* Age: > or = 18 years
* Ethnicity and race: All ethnic and racial backgrounds welcome
* Elevation of breath hydrogen after ingestion of 25 g of lactose > 20 ppm over baseline
* Planning to be available for clinic visits for the 6 weeks of study participation
* Ability and willingness to give written informed consent
* No known active psychiatric illness.

Exclusion Criteria:

* Intake of antibiotics or other medications within the past month
* History of diarrheal illness within past month
* Secondary lactase deficiency
* Self reported personal history of:

  *gastrointestinal conditions other than related with lactose maldigestion (IBS, IRB, Short bowel, malabsorption, celiac disease, GI surgery)
* Pregnant or Lactating
* Inability to communicate effectively with study personnel
* Protein allergy related to cow 's milk proteins or soybean proteins

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-02; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Change in Area Under the Curve (AUC) of Hydrogen (H2) production from day 1 at day 8 | Day 1 and day 8 of each milk phase
  Calculated as the H2 AUC above baseline at day 8 minus the H2 AUC above baseline at day 1 of each milk phase

SECONDARY OUTCOMES:
Severity of symptoms of lactose intolerance for each milk phase | Day 7 of each milk phase
  A validated gastrointestinal symptom log was used to mark on a 10-cm visual analog scale of 0 to 10 the severity of 4 symptoms: flatulence/gas, diarrhea, audible bowel sounds, and abdominal cramping.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Gardner, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mummah S, Oelrich B, Hope J, Vu Q, Gardner CD. Effect of raw milk on lactose intolerance: a randomized controlled pilot study. Ann Fam Med. 2014 Mar-Apr;12(2):134-41. doi: 10.1370/afm.1618. PMID 24615309
- See also: Study description and summary of results — https://med.stanford.edu/nutrition/research/completed-studies/raw-milk-study.html